CLINICAL TRIAL: NCT04133727
Title: Suiting up to Teach Pharmacy Students Empathy
Brief Title: Suiting up to Empathy
Acronym: PHARMSIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Associate Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHARMSIM
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Empathy
Keywords: randomised; simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will wear a simulation suit in which will mimic the physical limitations experienced by older adults. In addition, they will participate in a polypharmacy workshop which allows them to communicate with older adults
  Interventions: Behavioral: Use of an ageing suit
- Control (Active Comparator): This group will participate in a polypharmacy workshop which allows them to communicate with older adults
  Interventions: Other: Polypharmacy workshop

INTERVENTIONS:
Behavioral: Use of an ageing suit — The simulation suit consists of a pair glasses which simulates narrowing of visual field; a pair of gloves ; a vest ; elbow and knee wraps and sand bags worn on the wrists and ankles
  Other Names: PAUL Simulation Suit
  Arms: Intervention
Other: Polypharmacy workshop — Participants will conduct a full medication review for older adults within 1 hour and develop a medication list which can be used for counselling of older adults
  Other Names: Medication review polypharmacy workshop
  Arms: Control

SUMMARY:
Healthcare professionals with a positive attitude and empathetic towards older adults are at a better position to deliver quality healthcare. In this study, the investigators randomized pharmacy students to either a polypharmacy workshop or an immersive aging simulation suit and polypharmacy workshop to examine if simulation will enhance empathy levels among students

DETAILED DESCRIPTION:
Healthcare professionals with a positive attitude and empathetic towards older adults are at a better position to deliver quality healthcare. In this study, the investigators randomized pharmacy students to either a polypharmacy workshop or an immersive aging simulation suit and polypharmacy workshop to examine if simulation will enhance empathy levels among students. This will be performed in all year 1 pharmacy students

ELIGIBILITY:
Inclusion Criteria:

* All pharmacy students enrolled in the Pharmacy program

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Jefferson Empathy Scale | Baseline at Week 0 to Post Workshop at Week 12
  Change in empathy

SECONDARY OUTCOMES:
Subjective global question seeking opinion on the workshop and activity | Post intervention at Week 12
  Open ended qualitative response

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Lee, Principal Investigator — Monash University
Locations (1):
- Shaun Lee, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD can be requested from PI upon reasonable request

REFERENCES:
- [Derived] Lee SWH, Teh PL. "Suiting Up" to Enhance Empathy Toward Aging: A Randomized Controlled Study. Front Public Health. 2020 Aug 25;8:376. doi: 10.3389/fpubh.2020.00376. eCollection 2020. PMID 32984232